CLINICAL TRIAL: NCT01806129
Title: EROS: Engendering Reproductive Health Within Oncologic Survivorship
Brief Title: Reproductive Health Program in Patients With Cancer
Acronym: EROS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ECOG-ACRIN Cancer Research Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: Eastern Cooperative Oncology Group (Network)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: E1Q11; NCI-2012-02869 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); U10CA037403 (NIH)
Record Dates: First submitted 2013-02-19; First posted 2013-03-07 (Estimated); Results first posted 2022-10-05 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-02

CONDITIONS: Malignant Neoplasm
Keywords: reproductive health
MeSH Terms: conditions — Neoplasms | interventions — Algorithms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (no intervention) (Active Comparator): Patients undergo usual standard practice related to reproductive health.
  Interventions: Other: Standard practice related to reproductive heath
- Arm B (reproductive health program) (Experimental): Patients undergo reproductive health program comprising didactics, reproductive health assessment and navigating algorithm, and network development.
  Interventions: Other: Training modules, algorithm, referral development

INTERVENTIONS:
Other: Standard practice related to reproductive heath — Patients undergo usual standard practice related to reproductive health.
  Arms: Arm A (no intervention)
Other: Training modules, algorithm, referral development — Patients undergo reproductive health program comprising didactics, reproductive health assessment and navigating algorithm, and network development.
  Arms: Arm B (reproductive health program)

SUMMARY:
This clinical trial studies reproductive health program in patients with cancer. A reproductive health program may improve patients' understanding of reproductive risks and receipt of appropriate treatment to achieve their reproductive health goals.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the success of the implementation of reproductive health programming (Didactics, Engendering Reproductive Health Within Oncologic Survivorship [EROS] Reproductive Health Assessment and EROS Trial Algorithm) among reproductive aged females (15-55) with cancer.

SECONDARY OBJECTIVES:

I. To assess the degree of discrepancy between patients and their clinicians in estimates of significance of the reproductive health goals for the patient.

II. To evaluate baseline and follow-up reproductive health assessments for trends in reproductive health choices relating to oncofertility, oncocontraception and pregnancy over the 2-year study period.

III. To identify clinical and demographic factors that predict the adequacy of reproductive health care management.

TERTIARY OBJECTIVES:

I. To perform a longitudinal study following endocrine markers of fertility in a cohort of the first 200 registered EROS trial patients who agree to participate.

II. To perform a longitudinal study of sexual function using the Patient-Reported Outcomes Measurement Information System (PROMIS) sexual function survey in all subjects participating in the EROS Trial.

OUTLINE: Participating institutions are randomized to 1 of 2 arms. Patients are assigned to a study arm depending on the institutional assignment.

ARM A: Patients undergo usual standard practice related to reproductive health. ARM B: Patients undergo reproductive health program comprising didactics, reproductive health assessment and navigating algorithm, and network development.

After completion of study intervention, patients are followed up periodically.

ELIGIBILITY:
Inclusion Criteria:

* Female patients presenting with initial diagnosis of any type of cancer, including patients with ductal carcinoma in situ (DCIS)
* Pre-menopausal patients within the reproductive age range of 15-55 years; pre-menopausal is defined as females meeting the following criteria:

  * Patients not currently on hormonal contraception with the presence of menses in the past 6 months
  * If no menstruation in the past 6 months, without hormonal manipulation, then confirmed follicle-stimulating hormone (FSH) < 23mlU/mL
  * If age < 47 years and on hormonal contraception, then patient will be eligible regardless of menstrual history
  * If age ≥ 47 years and on hormonal contraception, then FSH confirmed < 23mIU/mL
* Pregnant women are eligible to participate in this study
* Patients must have the cognitive ability to participate in the study

Exclusion Criteria:

* Patients who have initiated chemotherapy, radiation therapy or endocrine therapy prior to registration to this study
* Prior hysterectomy, bilateral oophorectomy or sterilization of any method

Ages: 15 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 434 (Actual)
Dates: Start 2016-09-02 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2025-12-30 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Ashlesha Patel, Principal Investigator — Eastern Cooperative Oncology Group
Locations (109):
- United States (109):
  - Baptist Memorial Hospital and Fowler Family Cancer Center - Jonesboro, Jonesboro, Arkansas
  - Rocky Mountain Cancer Centers-Aurora, Aurora, Colorado
  - Rocky Mountain Cancer Centers-Boulder, Boulder, Colorado
  - Cancer Center of Colorado at Sloan's Lake, Denver, Colorado
  - Rocky Mountain Cancer Centers-Sky Ridge, Lone Tree, Colorado
  - SCL Health Lutheran Medical Center, Wheat Ridge, Colorado
  - Augusta University Medical Center, Augusta, Georgia
  - John B Amos Cancer Center, Columbus, Georgia
  - Hawaii Cancer Care Inc-POB II, Honolulu, Hawaii
  - Queen's Cancer Cenrer - POB I, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Queen's Cancer Center - Kuakini, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Tripler Army Medical Center, Honolulu, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - John H Stroger Jr Hospital of Cook County, Chicago, Illinois
  - Carle on Vermilion, Danville, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - Medical Oncology and Hematology Associates-West Des Moines, Clive, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - Greater Regional Medical Center, Creston, Iowa
  - Medical Oncology and Hematology Associates-Laurel, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - Saint Joseph Hospital East, Lexington, Kentucky
  - Saint Joseph London, London, Kentucky
  - Ochsner LSU Health Monroe Medical Center, Monroe, Louisiana
  - LSU Health Sciences Center at Shreveport, Shreveport, Louisiana
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Health Partners Inc, Minneapolis, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Baptist Memorial Hospital and Cancer Center-Oxford, Oxford, Mississippi
  - CHI Health Saint Francis, Grand Island, Nebraska
  - OptumCare Cancer Care at Seven Hills, Henderson, Nevada
  - OptumCare Cancer Care at Oakey, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-San Martin, Las Vegas, Nevada
  - Ann M Wierman MD LTD, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Tenaya, Las Vegas, Nevada
  - OptumCare Cancer Care at Fort Apache, Las Vegas, Nevada
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Memorial Medical Center - Las Cruces, Las Cruces, New Mexico
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - Montefiore Medical Center-Weiler Hospital, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Strecker Cancer Center-Belpre, Belpre, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Columbus Oncology and Hematology Associates Inc, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Providence Cancer Institute Clackamas Clinic, Clackamas, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Paoli Memorial Hospital, Paoli, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - AnMed Health Cancer Center, Anderson, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Gibbs Cancer Center-Pelham, Greer, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Baptist Memorial Hospital and Cancer Center-Memphis, Memphis, Tennessee
  - Meharry Medical College, Nashville, Tennessee
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - MultiCare Auburn Medical Center, Auburn, Washington
  - MultiCare Gig Harbor Medical Park, Gig Harbor, Washington
  - MultiCare Good Samaritan Hospital, Puyallup, Washington
  - MultiCare Tacoma General Hospital, Tacoma, Washington
  - Aurora Cancer Care-Southern Lakes VLCC, Burlington, Wisconsin
  - Aurora Health Center-Fond du Lac, Fond du Lac, Wisconsin
  - Aurora Cancer Care-Grafton, Grafton, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Aurora Cancer Care-Kenosha South, Kenosha, Wisconsin
  - Aurora Cancer Care-Milwaukee, Milwaukee, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic-Two Rivers, Two Rivers, Wisconsin
  - Aurora Cancer Care-Milwaukee West, Wauwatosa, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
  - Cheyenne Regional Medical Center-West, Cheyenne, Wyoming

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data may be made available upon request as per the ECOG-ACRIN Data Sharing Policy.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was activated on September 30, 2015 for site start-up preparation, opened to accrual on July 14, 2016, accrued its first patient on September 2, 2016, and closed to accrual on April 28, 2021 with a total of 434 patients accrued by 17 NCI Community Oncology Research Program (NCORP) sites.
Period: Overall Study
Arm/Group | Arm A (no Intervention) | Arm B (Reproductive Health Program)
Started | 278 | 156
Eligible and Analyzable Patients | 269 | 151
Completed | 278 | 156
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Only eligible patients were included in this analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A (no Intervention) | Arm B (Reproductive Health Program) | Total
Number analyzed (Participants) | 269 | 151 | 420
Age, Continuous [Median (Full Range); unit: years] | 41 [19 to 55] | 39 [18 to 54] | 41 [18 to 55]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 269 | 151 | 420
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 27 | 40 | 67
  Not Hispanic or Latino | 229 | 108 | 337
  Unknown or Not Reported | 13 | 3 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 24 | 5 | 29
  Native Hawaiian or Other Pacific Islander | 7 | 1 | 8
  Black or African American | 56 | 26 | 82
  White | 148 | 114 | 262
  More than one race | 3 | 0 | 3
  Unknown or Not Reported | 31 | 4 | 35

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients With Appropriate Reproductive Health Management
Description: Appropriate reproductive health management was determined using the followings: (1) Females that were pregnant or interested in immediate pregnancy (defined as within 1 year of enrollment) were given referral to obstetrician/gynecologist or counseled about pregnancy options (2) Females interested in future childbearing were counseled or given a referral for fertility preservation if requested (3) Females who were not interested in immediate pregnancy were given a referral or counseling to select family planning that was consistent with plans for sexual activity and future childbearing. If a female fell into category 1, 2, or 3, and the appropriate referral occurred within 3 months of enrollment, then appropriate reproductive health management was achieved. For patients with appropriate reproductive health management in place before the baseline visit, they were included in the analysis and counted as having appropriate reproductive health management.
Time Frame: At baseline and 3 months
Population: Only eligible patients who were evaluable for the primary endpoint were included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (no Intervention) | Arm B (Reproductive Health Program)
Number analyzed (Participants) | 245 | 134
Participants
  Without appropriate reproductive health management | 129 | 46
  With appropriate reproductive health management | 116 | 88
Statistical Analysis 1: Comparison: Arm A (no Intervention) vs Arm B (Reproductive Health Program); Test type: Superiority; Odds Ratio (OR) = 2.07, 90% CI 2-sided [1.29 to 3.31] — Odds ratio represents the odds of adopting the appropriate reproductive health management for patients with intervention compared to the odds among patients without intervention. Odds ratio was calculated by GEE analysis

2. Secondary Outcome: Difference in Rating Between Patients and Their Clinicians in Importance of Fertility Maintenance
Description: The rating on the importance of fertility maintenance was assessed among patients and the corresponding treating physicians. The rating scale ranges between 1 and 10. Higher scores indicate more importance of fertility maintenance. The difference in rating was calculated by subtracting patient rating from physician's rating.
Time Frame: At baseline
Population: Patients with both patient rating and physician rating available were included in this analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm A (no Intervention) | Arm B (Reproductive Health Program)
Number analyzed (Participants) | 260 | 145
score on a scale | 0.03 (0.67) | 0.12 (0.67)

3. Secondary Outcome: The Changes in Reproductive Health Status From Baseline to 3 Months
Description: Patient's reproductive health choices relating to oncofertility, oncocontraception and pregnancy was assessed at baseline and 3 months. Patient's reproductive health status is categorized into the following categories:
  * Sextually active & childbearing not completed
  * Sextually active & childbearing completed
  * Sextually not active & childbearing not completed
  * Sextually not active & childbearing completed
  * Sexuality unknown & childbearing not completed
  * Sexuality unknown & childbearing completed
  * Pregnant/Pregnancy in 1 year
  * Missing/Unknown
Time Frame: Baseline and 3 months
Population: All eligible/analyzable patients were included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (no Intervention) | Arm B (Reproductive Health Program)
Number analyzed (Participants) | 269 | 151
Participants
  Baseline: Sextually active & childbearing not completed at 3 months | 52 | 34
  Baseline: Sextually active & childbearing completed at 3 months | 109 | 58
  Baseline: Sextually not active & childbearing not completed at 3 months | 32 | 20
  Baseline: Sextually not active & childbearing completed at 3 months | 62 | 35
  Baseline: Sexuality unknown & childbearing not completed at 3 months | 2 | 0
  Baseline: Sexuality unknown & childbearing completed at 3 months | 3 | 0
  Baseline: Pregnant/Pregnancy in 1 year at 3 months | 9 | 4
  Baseline: Missing/Unknown at 3 months | 0 | 0
  3 months: Sextually active & childbearing not completed at 3 months | 37 | 14
  3 months: Sextually active & childbearing completed at 3 months | 88 | 45
  3 months: Sextually not active & childbearing not completed at 3 months | 20 | 10
  3 months: Sextually not active & childbearing completed at 3 months | 71 | 37
  3 months: Sexuality unknown & childbearing not completed at 3 months | 0 | 0
  3 months: Sexuality unknown & childbearing completed at 3 months | 2 | 2
  3 months: Pregnant/Pregnancy in 1 year at 3 months | 18 | 15
  3 months: Missing/Unknown at 3 months | 33 | 28

4. Secondary Outcome: Associations Between Clinical and Demographic Factors and Adequacy of Reproductive Health Care Management
Description: as for outcome 1
Time Frame: Baseline and 3 months
Population: Eligible patients with primary endpoint evaluated were included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (no Intervention) | Arm B (Reproductive Health Program)
Number analyzed (Participants) | 245 | 134
Participants
  Completed childbearing at baseline: number analyzed (Participants) | 159 | 83
  Completed childbearing at baseline: With appropriate reproductive health management | 79 | 62
  Completed childbearing at baseline: Without appropriate reproductive health management | 80 | 21
  Childbearing not completed at baseline: number analyzed (Participants) | 86 | 51
  Childbearing not completed at baseline: With appropriate reproductive health management | 37 | 26
  Childbearing not completed at baseline: Without appropriate reproductive health management | 49 | 25

5. Other Pre Specified Outcome: Levels of Endocrine Markers of Fertility
Description: Reproductive health-related biomarkers, including follicle-stimulating hormone (FSH), anti-müllerian hormone (AMH), thyroid stimulating hormone (TSH) and Thyroid peroxidase (TPO), were evaluated through blood samples collected at baseline and 3, 6, 12, 24 months.
Time Frame: Baseline and 3, 6, 12, 24 months
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Sexual Function Score by Patient-Reported Outcomes Measurement Information System (PROMIS)
Description: Sexual function was evaluated using PROMIS sexual function survey brief profile V1.0. All subdomain scores (except for the orgasm subdomain) are expressed as T-scores with a mean of 50 and a standard deviation of 10. A raw summed score is created for each domain. For Global Satisfaction with Sex Life, the raw summed score can range from 2 (endorsed "Not at all" to both items) to 10 (endorsed "Very" or "Very much" to both items). Higher scores indicate more satisfaction/interest/lubrication/discomfort/ability with sex life. Lower scores indicate less satisfaction/interest/lubrication/discomfort/ability with sex life.
Time Frame: Baseline and 3, 6, 12, 24 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed.
Description: Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed.
Arm/Group | Arm A (no Intervention) | Arm B (Reproductive Health Program)
All-Cause Mortality (participants affected / at risk) | 10/278 | 7/156
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-17): https://cdn.clinicaltrials.gov/large-docs/29/NCT01806129/Prot_SAP_000.pdf